CLINICAL TRIAL: NCT01922622
Title: Determination of the Initial Minimum Effective Dose of 0.5% Bupivacaine With 20mcg of Fentanyl Via a Spinal Catheter for Operative Fixation of Fractured Neck of Femur.
Brief Title: Minimum Effective Intrathecal Dose of Local Anaesthetic With Fentanyl for Fractured Neck of Femur(Dose Finding Study).
Status: Completed | Type: Observational
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, tomas hitka, Clinical fellow in Regional Anaesthesia, Cork University Hospital
Other Study IDs: ECM 4(qqqq)07/05/13
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Minimum Effective Dose of Local Anaesthetic With Fentanyl
Keywords: minimum effective dose of local anaesthetic; spinal catheter; fractured neck of femur; a step up, step down methodology
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bipolar hemiarthroplasty.: Group of patients who will stay in lateral position during whole surgery.
- Dynamic hip screw.: Group of patients who will be supine during surgery.

SUMMARY:
Fractured neck of femur (FNF) is a common cause of admission to hospital in elderly patients with multiple comorbidities. Anaesthetic management of this patient group is extremely challenging.Neuraxial anaesthesia with minimum doses of local anaesthetic agents administered via a spinal catheter leads to better cardiovascular stability.The minimum dose of local anaesthetic with intrathecal fentanyl was not established yet.We propose to study and determine the initial minimum local anaesthetic dose (MLAD) of 0.5% bupivacaine with 20 mcg of fentanyl administered via a spinal catheter to achieve a sensory block up to T10 for the operative fixation of FNF.We will use a previously well established Dixon and Massey "up-and-down method" to calculate initial MLAD in this prospective, observational trial.

Objectives: We would like to determine the initial MLAD of 0.5% bupivacaine with 20mcg of fentanyl administered via a spinal catheter required to achieve a sensory block up to T10 on the side of FNF.

Outcomes

Primary outcome:

1. Initial MLAD of 0.5% bupivacaine with 20mcg of fentanyl required for a sensory block up to T10 on the side of FNF.

   Secondary outcomes:
2. Total dose of 0.5% bupivacaine with 20mcg of fentanyl required for the operative fixation of fractured neck of femur.
3. The effect on haemodynamic variables (blood pressure, heart rate).
4. Incidence of side effects
5. The length of postoperative analgesia (the time from the last dose of local anaesthetic administered intrathecally to VAS>3).
6. The time to first rescue analgesic requirement

Study Design Prospective, observational trial.

Study Size Based on the previously well established Dixon and Massey "up-and-down method"(10), we will recruit patients until a successful spinal block has been achieved in six consecutive patients who received a specific dose. This is the requirement to calculate the initial MLAD.

ELIGIBILITY:
Inclusion Criteria:

* fractured neck of femur
* Above 60 years
* American Society of Anesthetists(ASA) I to III

Exclusion Criteria:

* Patient refusal
* Outside Age Range
* Contraindications to spinal anaesthesia
* Head injury or other associated injuries
* Loss of consciousness and signs of acute coronary syndrome
* Mini-Mental Score < 25 (Appendix 2)
* Allergy to bupivacaine, lignocaine or fentanyl

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with fractured neck of femur undergoing surgical repair of their fracture
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Initial MLAD of 0.5% bupivacaine with 20mcg of fentanyl required for a sensory block up to T10 on the side of FNF | 15min
  A blinded observer will assess the dermatome level of sensory blockade with an ice-cold test (ethyl-chloride spray) bilaterally after the injection of the local anaesthetic. Block assessment will be performed every 5min up to 15 min after completion of the initial intrathecal injection. Sensory block up to T10=positive result Sensory block below T10=negative result.

SECONDARY OUTCOMES:
Total dose of 0.5% bupivacaine with 20mcg of fentanyl required for the operative fixation of fractured neck of femur | Duration of surgery.
  Initial dose and all top ups will be recorded and analysed in conjunction with the length of surgery and surgical procedure used to fix FNF.
The effect on haemodynamic variables (blood pressure, heart rate). | Duration of surgery.
  Noninvasive automated blood pressure and heart rate measurements will be recorded before the spinal anaesthesia (baseline) and every three minutes after the end of local anesthetic injection until the end of surgery.Hypotension is defined as a decrease of more than 20% from the baseline systolic arterial blood pressure (SAP). Severe hypotension is defined as a decrease in SAP more than 30% of baseline value. Hypotension will be treated with IV boluses of ephedrine 6 mg if the heart rate is below 60/minutes or phenylephrine 100 mcg if the heart rate is above 60/minutes.The number of hypotensive episodes, a total amount of vasopressor administered, and the i.v. fluid infused will be recorded as well as duration of anaesthesia.

OTHER OUTCOMES:
Incidence of side effects. | 24-48 hours
  Patients will be interviewed 24-48 hours after surgery regarding side effects of spinal anaesthesia (headache, pruritus,postoperative nausea and vomiting,urinary retention,neurological deficit)
The length of postoperative analgesia (the time from the last dose of local anaesthetic administered intrathecally to VAS>3). | 1-2 hours
  The time from the last top up of local anaesthetic to VAS >3 and to the first dose of break through analgesia will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hitka, RA fellow, Principal Investigator — Cork University Hospital; Gabriella Iohom, consultant, Study Chair — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

REFERENCES:
- [Background] Hocking G, Wildsmith JA. Intrathecal drug spread. Br J Anaesth. 2004 Oct;93(4):568-78. doi: 10.1093/bja/aeh204. Epub 2004 Jun 25. No abstract available. PMID 15220175
- [Background] Minville V, Fourcade O, Grousset D, Chassery C, Nguyen L, Asehnoune K, Colombani A, Goulmamine L, Samii K. Spinal anesthesia using single injection small-dose bupivacaine versus continuous catheter injection techniques for surgical repair of hip fracture in elderly patients. Anesth Analg. 2006 May;102(5):1559-63. doi: 10.1213/01.ane.0000218421.18723.cf. PMID 16632842
- [Background] Stocks GM, Hallworth SP, Fernando R, England AJ, Columb MO, Lyons G. Minimum local analgesic dose of intrathecal bupivacaine in labor and the effect of intrathecal fentanyl. Anesthesiology. 2001 Apr;94(4):593-8; discussion 5A. doi: 10.1097/00000542-200104000-00011. PMID 11379678
- [Background] Idowu OA, Sanusi AA, Eyelade OR. Effects of intrathecally administered fentanyl on duration of analgesia in patients undergoing spinal anaesthesia for elective caesarean section. Afr J Med Med Sci. 2011 Sep;40(3):213-9. PMID 22428515
- [Background] Sell A, Olkkola KT, Jalonen J, Aantaa R. Minimum effective local anaesthetic dose of isobaric levobupivacaine and ropivacaine administered via a spinal catheter for hip replacement surgery. Br J Anaesth. 2005 Feb;94(2):239-42. doi: 10.1093/bja/aei015. Epub 2004 Oct 29. PMID 15516345
- [Background] O'Donnell BD, Iohom G. An estimation of the minimum effective anesthetic volume of 2% lidocaine in ultrasound-guided axillary brachial plexus block. Anesthesiology. 2009 Jul;111(1):25-9. doi: 10.1097/ALN.0b013e3181a915c7. PMID 19512869
- [Background] Casati A, Baciarello M, Di Cianni S, Danelli G, De Marco G, Leone S, Rossi M, Fanelli G. Effects of ultrasound guidance on the minimum effective anaesthetic volume required to block the femoral nerve. Br J Anaesth. 2007 Jun;98(6):823-7. doi: 10.1093/bja/aem100. Epub 2007 May 3. PMID 17478453
- [Background] Hartwell BL, Aglio LS, Hauch MA, Datta S. Vertebral column length and spread of hyperbaric subarachnoid bupivacaine in the term parturient. Reg Anesth. 1991 Jan-Feb;16(1):17-9. PMID 2007099
- [Background] Egan TD, Kern SE, Muir KT, White J. Remifentanil by bolus injection: a safety, pharmacokinetic, pharmacodynamic, and age effect investigation in human volunteers. Br J Anaesth. 2004 Mar;92(3):335-43. doi: 10.1093/bja/aeh075. PMID 14970134
- [Background] Machata AM, Gonano C, Holzer A, Andel D, Spiss CK, Zimpfer M, Illievich UM. Awake nasotracheal fiberoptic intubation: patient comfort, intubating conditions, and hemodynamic stability during conscious sedation with remifentanil. Anesth Analg. 2003 Sep;97(3):904-908. doi: 10.1213/01.ANE.0000074089.39416.F1. PMID 12933427
- [Derived] Hitka T, O'Sullivan J, Szucs S, Iohom G. Determination of the initial minimum effective dose of 0.5% bupivacaine with 20 mug of fentanyl for an operative fixation of fractured neck of femur: a prospective, observational trial. Minerva Anestesiol. 2021 Jul;87(7):766-773. doi: 10.23736/S0375-9393.21.15012-6. Epub 2021 Feb 16. PMID 33591143